CLINICAL TRIAL: NCT02864680
Title: Electrophysiological Study of the Functioning of Magnocellular Visual Pathway in Regular Cannabis Users
Acronym: CAUSA MAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2013-A00097-38
Record Dates: First submitted 2016-08-03; First posted 2016-08-12 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2019-06

CONDITIONS: Cannabis Use
Keywords: cannabis; magnocellular pathway
MeSH Terms: conditions — Marijuana Abuse | interventions — Gene Expression; Succimer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cannabis users (Other)
  Interventions: Other: Electroretinography; Other: Contrast sensitivity test during Electroencephalography; Other: Visual simultaneity test during Electroencephalography; Other: Face perception test during Electroencephalography; Other: CAST (cannabis abuse screening test); Other: Delayed Matching to Sample (DMS) test; Other: Spatial Working Memory (SWM) test; Other: Rapid Visual Information Processing (RVP) test; Other: Test for attentional performance (TAP) / Divided Attention; Other: Collection of saliva sample
- Healthy volunteers, not cannabis/tobacco users (Other)
  Interventions: Other: Electroretinography; Other: Contrast sensitivity test during Electroencephalography; Other: Visual simultaneity test during Electroencephalography; Other: Face perception test during Electroencephalography; Other: Delayed Matching to Sample (DMS) test; Other: Spatial Working Memory (SWM) test; Other: Rapid Visual Information Processing (RVP) test; Other: Test for attentional performance (TAP) / Divided Attention; Other: Collection of saliva sample
- Healthy volunteers, tobacco users (Other)
  Interventions: Other: Electroretinography; Other: Contrast sensitivity test during Electroencephalography; Other: Visual simultaneity test during Electroencephalography; Other: Face perception test during Electroencephalography; Other: Delayed Matching to Sample (DMS) test; Other: Spatial Working Memory (SWM) test; Other: Rapid Visual Information Processing (RVP) test; Other: Test for attentional performance (TAP) / Divided Attention; Other: Collection of saliva sample
- Schizophrenia patients (Other)
  Interventions: Other: Electroretinography; Other: Contrast sensitivity test during Electroencephalography; Other: Visual simultaneity test during Electroencephalography; Other: Face perception test during Electroencephalography; Other: CAST (cannabis abuse screening test); Other: PANSS (Positive And Negative Symptoms Scale) test; Other: Delayed Matching to Sample (DMS) test; Other: Spatial Working Memory (SWM) test; Other: Rapid Visual Information Processing (RVP) test; Other: Test for attentional performance (TAP) / Divided Attention; Other: Collection of saliva sample

INTERVENTIONS:
Other: Electroretinography
Other: Contrast sensitivity test during Electroencephalography — Stimuli are black and white grids, having different range of spatial frequencies, presented with different contrasts on a grey background thanks to a computer monitor, in a dark room. Participants are requested to maintain central fixation. During the test patients stay sit, head hold by chin strap. A pause can be asked by participant and done at every moment. This test lasts approximately 30 minutes.
Other: Visual simultaneity test during Electroencephalography — Two vertical bars are showed on a monitor, on the link and right of point of central fixation. Bars appear simultaneously or with a 10 to 200 ms asynchrony. Participants must determine whether stimuli are simultaneous or asynchronous and answer pressing the link button for simultaneity or right button for asynchrony. During the test patients stay sit, head hold by chin strap. A pause can be asked by participant and done at every moment. This test lasts approximately 30 minutes.
Other: Face perception test during Electroencephalography — Faces filtered in different spatial frequence ranges are showed randomly on a monitor, in a dark room. Participants must maintain a central fixation thank to a fixation cross. During the test patients stay sit, head hold by chin strap. A pause can be asked by participant and done at every moment. This test lasts approximately 30 minutes.
Other: CAST (cannabis abuse screening test)
  Arms: Cannabis users; Schizophrenia patients
Other: PANSS (Positive And Negative Symptoms Scale) test
  Arms: Schizophrenia patients
Other: Delayed Matching to Sample (DMS) test
Other: Spatial Working Memory (SWM) test
Other: Rapid Visual Information Processing (RVP) test
Other: Test for attentional performance (TAP) / Divided Attention
Other: Collection of saliva sample — In case of specific consent of participant to ancillary study, for ancillary study

SUMMARY:
This study will evaluate the impact of regular use of cannabis on the spatial sensitivity of magnocellular system (visual event-related potential, visual ERP).

Secondary purposes of this study are to evaluate the impact of regular use of cannabis on the temporal sensitivity of magnocellular system (visual event-related potential), on the dynamics of cortical visual processing during face perception test (visual event-related potential) and on functioning of retinal photopic and scotopic systems (electroretinogram).

The ancillary study is a genetic analysis of a group of candidate genes that aims to identify biomarkers for changes in visual processing. This will allow to distinguish among more homogeneous and specific groups in future studies on larger cannabis user population. This ancillary study concerns all participants subject to their informed consent (facultative study).

ELIGIBILITY:
Inclusion Criteria:

* Affiliation to social security plan
* Normal visual acuity or adjusted to normal and normal dilated fundus examination
* Signature of informed consent
* Cannabis user group: More than 7 cannabis uses per week during the previous month
* Cannabis user group: Positive urinary analysis for presence of cannabis
* Healthy, non user control group: Absence of cannabis and tobacco use during last 12 months
* Healthy, non user control group: Negative urinary analysis for presence of cannabis
* Healthy, non user control group: Age and sex matching with cannabis user group
* Healthy, tobacco user control group: Tobacco use from at least 12 months
* Healthy, tobacco user control group: Low to very strong addiction to tobacco (Fagerström test)
* Healthy, tobacco user control group: Absence of cannabis use from more than 12 months
* Healthy, tobacco user control group: Negative urinary analysis for presence of cannabis
* Healthy, tobacco user control group:Age and sex matching with cannabis user group
* Schizophrenia patient control group: Schizophrenia according to DMS IV criteria (MINI test)
* Schizophrenia patient control group: Absence of cannabis use from more than one month (regardless of tobacco use)
* Schizophrenia patient control group: Negative urinary analysis for presence of cannabis
* Schizophrenia patient control group: Age and sex matching with cannabis user group

Exclusion Criteria:

* Acute psychiatric pathology (axis I of DSM IV, measured by MINI) except anxiety disorder (except schizophrenia group)
* Deficiency of the subject making difficult or impossible his/her participation to the study or the comprehension of the information
* Dyslexia
* Addiction to alcohol according to AUDIT scale
* Abuse or addiction to other substances according to DSM IV criteria
* Acute retinal disorder
* Chronic glaucoma
* Ophthalmic pathology affecting visual acuity
* Current ocular infection
* Persons under guardianship, curatorship or judicial protection
* Pregnant or breast-feeding women
* Persons with life-and-death emergency
* Absence of social security plan
* Results of preliminary medical examinations incompatible with the study
* Simultaneous participation to another therapeutic interventional study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 163 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Amplitude of P100 wave in contrast sensibility test | up to 1 month
Culmination time of the P100 wave in contrast sensibility test | up to 1 month

SECONDARY OUTCOMES:
Amplitude of P100 wave in visual simultaneity test | up to 1 month
Culmination time of P100 wave in visual simultaneity test | up to 1 month
Amplitude of P100 wave in face perception test | up to 1 month
Amplitude of N170 wave in face perception test | up to 1 month
Culmination time of P100 wave in face perception test | up to 1 month
Culmination time of N170 wave in face perception test | up to 1 month
Amplitude of "a" wave in different ERG sequences | day 0
Amplitude of "b" wave in different ERG sequences | day 0
Culmination time of "a" wave in different ERG sequences | day 0
Culmination time of "b" wave in different ERG sequences | day 0

OTHER OUTCOMES:
Relationship between variants of candidate genes for alterations of visual treatment and amplitude of P100 wave in contrast sensibility test | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Vincent LAPREVOTE, Principal Investigator — Maison des Addictions - CHU de Nancy, France
Locations (1):
- Maison des Addictions - CHU de Nancy, Hôpital St Julien, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Remy I, Bernardin F, Ligier F, Krieg J, Maillard L, Schwan R, Schwitzer T, Laprevote V. Association between retinal and cortical visual electrophysiological impairments in schizophrenia. J Psychiatry Neurosci. 2023 May 19;48(3):E171-E178. doi: 10.1503/jpn.220224. Print 2023 May-Jun. PMID 37208126
- [Derived] Bernardin F, Schwitzer T, Schwan R, Angioi-Duprez K, Ligier F, Bourion-Bedes S, Jansen C, Giersch A, Laprevote V. Altered central vision and amacrine cells dysfunction as marker of hypodopaminergic activity in treated patients with schizophrenia. Schizophr Res. 2022 Jan;239:134-141. doi: 10.1016/j.schres.2021.11.049. Epub 2021 Dec 7. PMID 34891077
- [Derived] Remy I, Schwitzer T, Albuisson E, Schwan R, Krieg J, Bernardin F, Ligier F, Lalanne L, Maillard L, Laprevote V. Impaired P100 among regular cannabis users in response to magnocellular biased visual stimuli. Prog Neuropsychopharmacol Biol Psychiatry. 2022 Mar 8;113:110437. doi: 10.1016/j.pnpbp.2021.110437. Epub 2021 Sep 11. PMID 34520807